CLINICAL TRIAL: NCT04829773
Title: An Open-Label Study Evaluating the Effect of Food on the Pharmacokinetics of Palovarotene and the Effect of Palovarotene on the Pharmacokinetics of the CYP3A4 Substrate Midazolam in Two Cohorts of Healthy Adult Subjects
Brief Title: Study Evaluating the Effect of Food on the Pharmacokinetics of Palovarotene and the Effect of Palovarotene on the Pharmacokinetics of the CYP3A4 Substrate Midazolam in Two Cohorts of Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PVO-1A-102
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Fibrodysplasia Ossificans Progressiva
MeSH Terms: conditions — Myositis Ossificans | interventions — Palovarotene; Midazolam

STUDY DESIGN:
Intervention Model Description: This study had two components. One component evaluated the effect of food and the effect of swallowing capsule whole versus sprinkling on apple sauce on the PK/bioavailability of palovarotene, and the other component evaluated the effect of palovarotene on the PK of the CYP3A4 substrate midazolam. The PK of palovarotene after single and multiple doses was also evaluated as part of the DDI component. Two cohorts of healthy adult subjects were enrolled, one for each component.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PK Cohort 1 (Experimental): Subjects received three single oral doses of palovarotene on Days 1, 6, and 11, separated by 5-day washout periods.
  Sequence A-B-C: Subjects received a single oral dose of palovarotene whole capsule under fasting conditions (at least a 10-hour overnight fast); followed by a single oral dose of palovarotene whole capsule 30 minutes after the start of a standardized high-fat, high-caloric breakfast; and then followed by a single oral dose of palovarotene sprinkled on 1 teaspoon of apple sauce, administered 30 minutes after the start of a standardized high-fat, high-caloric breakfast.
  Interventions: Drug: Palovarotene
- PK Cohort 2 (Experimental): Subjects received three single oral doses of palovarotene on Days 1, 6, and 11, separated by 5-day washout periods.
  Sequence B-C-A: Subjects received a single oral dose of palovarotene whole capsule 30 minutes after the start of a standardized high-fat, high-caloric breakfast; followed by a single oral dose of palovarotene sprinkled on 1 teaspoon of apple sauce, administered 30 minutes after the start of a standardized high-fat, high-caloric breakfast; and then followed by a single oral dose of palovarotene whole capsule under fasting conditions (at least a 10-hour overnight fast).
  Interventions: Drug: Palovarotene
- PK Cohort 3 (Experimental): Subjects received three single oral doses of palovarotene on Days 1, 6, and 11, separated by 5-day washout periods.
  Sequence C-A-B: Subjects received a single oral dose of palovarotene sprinkled on 1 teaspoon of apple sauce, administered 30 minutes after the start of a standardized high-fat, high-caloric breakfast; followed by a single oral dose of palovarotene whole capsule under fasting conditions (at least a 10-hour overnight fast); and then followed by a single oral dose of palovarotene whole capsule 30 minutes after the start of a standardized high-fat, high-caloric breakfast.
  Interventions: Drug: Palovarotene
- Drug-Drug interaction (DDI) Cohort (Experimental): On the morning of Day 1, subjects received a single dose of midazolam 30 minutes after the start of a standardized breakfast. On Day 2 (after the 24-hour midazolam blood draw) through Day 15, subjects received a daily, single dose of palovarotene in the morning 30 minutes after the start of a standardized breakfast. A second dose of midazolam was administered on Day 15 in the morning (immediately following the palovarotene dose) 30 minutes after the start of a standardized breakfast.
  Interventions: Drug: Palovarotene; Drug: midazolam

INTERVENTIONS:
Drug: Palovarotene — oral capsules
Drug: midazolam — oral syrup
  Arms: Drug-Drug interaction (DDI) Cohort

SUMMARY:
Study to evaluate the effect of food and the effect of swallowing capsule whole versus sprinkling on apple sauce on the pharmacokinetics (PK)/bioavailability of palovarotene, and evaluate the effect of palovarotene on the PK of the CYP3A4 substrate midazolam.

ELIGIBILITY:
Key Inclusion Criteria:

* Generally healthy male or female aged 18 to 55 years, inclusive; body mass index (BMI) of 18 to 30 kg/m2 and a body weight of >50 kg; resting pulse of >45 bpm and <100 bpm; systolic and diastolic blood pressure of <140/90 mmHg

Key Exclusion Criteria:

* a history or current evidence of a clinically significant or uncontrolled disease, disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* exposure to synthetic oral retinoids or creams containing retinoids in the past 30 days prior to the signature of the informed consent.
* history or presence of silent infections, including positive tests for human immunodeficiency virus type 1 (HIV-1), human immunodeficiency virus type 2 (HIV-2), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* history of allergy or hypersensitivity to retinoids, gelatin, or lactose
* For the DDI component only, the subject had a history of allergy or hypersensitivity to benzodiazepines, midazolam, cherries, or midazolam formulation excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) observed plasma drug concentration | Days 1, 2, 3, 6, 7, 8, 11, 12, 13.
Time to reach maximum (peak) (t max) observed plasma concentration following drug administration | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
Area under the plasma concentration time (AUC 0-last) curve from time zero to the last quantifiable time point, calculated by linear-log trapezoidal summation | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
Area under the plasma concentration time curve from time zero to infinity (AUC 0-infinity) | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
  calculated by linear-log trapezoidal summation and extrapolated to infinity by addition of the last quantifiable plasma concentration divided by the elimination rate constant
Apparent terminal disposition rate constant/terminal rate constant yz | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
  determined by linear regression of the terminal points of the log-linear plasma concentration-time curve
Apparent terminal elimination half-life (t1/2) | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
Apparent volume of distribution after oral administration (Vd/F) | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
Apparent total clearance of the drug from plasma after oral administration (cLF) | Days 1, 2, 3, 6, 7, 8, 11, 12, 13
Area under the plasma concentration time curve from time zero to 24 hours only for DDI cohort | Days 1, 2, 15, 16
The last concentration before the next study drug administration at steady state for DDI cohort | Days 1, 2, 15, 16
Maximum (peak) observed plasma drug concentration at steady state for DDI cohort | Days 1, 2, 15, 16
Time to reach maximum (peak) observed plasma concentration following drug administration at steady state for DDI cohort | Days 1, 2, 15, 16
Minimum observed plasma concentration at steady state, taken as the lowest plasma concentration during dosing interval for DDI cohort | Days 1, 2, 15, 16
Accumulation ratio for DDI cohort | Days 1, 2, 15, 16

SECONDARY OUTCOMES:
Occurrence of Adverse Events (AEs) | from baseline until the end of study (16 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Cambridge Ipsen US, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Marino R, Dube L, Ogier J, Le Quan Sang KH. The Pharmacokinetic Profile of Palovarotene: An Open-Label Phase I Trial Investigating the Effect of Food and Potential for Drug-Drug Interaction in Healthy Participants. Eur J Drug Metab Pharmacokinet. 2023 Nov;48(6):691-707. doi: 10.1007/s13318-023-00856-2. Epub 2023 Oct 7. PMID 37804430